CLINICAL TRIAL: NCT05004857
Title: The Effect of Reading Therapy on Newborns
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Saul's Light Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-611
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Autonomic Nervous System Diseases
Keywords: Reading; Neonates; New borns; Autonomic nervous system
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patient arm (Experimental): The subject population will be newborn infants admitted to the Newborn Nursery (NN) at Tulane Lakeside Hospital. The investigators are anticipating some mothers can be recruited from the prenatal clinics who expect to deliver at Tulane Hospital during pregnancy as well.
  Interventions: Behavioral: Book reading

INTERVENTIONS:
Behavioral: Book reading — Prior to the first session, a research assistant will place electrodes on the infant and mother so that they study team can gather autonomic nervous system (ANS) response (sympathetic and parasympathetic) non-invasively using MindWare Portable Lab System (MindWare Technologies, Gahanna, Ohio). These electrodes will remain on the infant and mother throughout each session and be removed via adhesive removing pads following each session's data collection. This will minimize discomfort to both parties secondary to electrode removal and minimize risk of skin irritation by leaving electrodes in place for a prolonged period of time. Additional observational data before and after the reading sessions will be collected by the research assistant, including but not limited to: where the session is conducted (mother's arms, bassinet), activity level, vital signs, and any other observed behaviors throughout the session.

SUMMARY:
The primary purpose of this pilot study is to specifically examine the effect of parental reading on the ANS of mother and neonate in the hospital setting. The investigators will examine the effect of live maternal-infant reading on typically developing infants to better understand the physiological benefits of live reading on newborns.

DETAILED DESCRIPTION:
Supporting infant ANS development has been implicated in their improved cardiorespiratory and neuropsychiatric outcome; furthermore, improved parasympathetic activity, a branch of ANS, is a predictor of the mother-infant relationship, and the best marker for caregiving behavior. In Feldman and Eidelman's 2003 study, they demonstrated that mother-infant skin-to-skin contact, also known as Kangaroo Care, accelerates ANS maturation in pre-term infants, which is critical for their recovery. If reading is shown to have a positive effect on mother infant ANS, hospitals will be able to incorporate this into practice as a feasible alternative for when Kangaroo Care isn't possible. The investigators hope to learn if these reading interventions will help to mitigate distress symptoms, among both mother and baby, within the hospital. The investigators will examine the association of reading therapy with the infant's crying patterns, length of stay in the hospital, weight gain, and behavior compared to before the reading was done.

Seeing that Scala's findings from 2018 is the only indication of physiologic benefits of reading to infants in the hospital, additional research is required in this particular area. The testing and application of reading therapy in the Neonatal Intensive Care Unit (NICU) would improve a high-stress environment for both parents and infants. Data collected from this project will not only add some much-needed information to the limited knowledge of the physiological effects of reading on neonates, but also demonstrate how infant outcomes can be improved in a cost-effective, efficient manner within the hospital setting.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Tulane-Lakeside Hospital Newborn Nursery
* Corrected gestational age 34 weeks or older
* No identified hearing disorder
* Do not have a diagnosed developmental disability (i.e. Down Syndrome)
* Do not have Fetal Alcohol Syndrome
* Medically cleared to participate in the study
* Biological mother able/willing to give consent in English & complete surveys.

Exclusion Criteria:

* Corrected gestational age < 34 weeks old
* Has an identified or potential hearing disorder (i.e, failed hearing screen)
* Has diagnosed developmental disability (i.e. Down syndrome)
* Has Fetal Alcohol Syndrome
* Is not medically cleared to participate in the study
* Biological mother unable/unwilling to give consent.

Ages: 1 Minute to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the change in vagal tone | 20 minutes of reading
  The change in vagal tone from the reading therapy will be measured using MindWare System, where an increase in vagal tone shows positive physiological outcomes in the newborns and mothers.
Determine the change in parasympathetic nervous system response | 20 minutes of reading
  The change in parasympathetic nervous system response from the reading therapy will be measured using MindWare System, where an increase in parasympathetic nervous system response shows positive physiological outcomes in the newborns and mothers.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Howell, MD, MS, Principal Investigator — Tulane University
Locations (1):
- Tulane University Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided